CLINICAL TRIAL: NCT07351253
Title: Analgeisc Effect of Erector Spinae Plane Block Versus Lateral Transversus Abdominis Plane Block in Patients Undergoing Open Abendectomy Surgery: a Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block Versus Lateral Transversus Abdominis Plane Block for Open Abendectomy Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-320-2024
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Appendicectomy; Postoperative Analgesia; Regional Anaesthesia
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP group (Active Comparator)
  Interventions: Other: Erector Spinae Plane Block
- TAP group (Active Comparator)
  Interventions: Other: Transversus abdominis plane (TAP) block

INTERVENTIONS:
Other: Erector Spinae Plane Block — Patients will receive the ESP block at the level of the 10th thoracic (T10) transverse process using a linear 6-13 MHz ultrasound transducer. A 20 mL of 0.25% bupivacaine will be injected below the muscle
  Arms: ESP group
Other: Transversus abdominis plane (TAP) block — Patient will received TAP block using the lateral approach while in supine position. A 20 mL of 0.25% bupivacaine will be injected after negative aspiration.
  Arms: TAP group

SUMMARY:
this aim of this study is to compare the analgesic effect of Erector spinae plane (ESP) block and lateral transversus abdominis plan (TAP) block in patients undergoing open appendectomy.

DETAILED DESCRIPTION:
regional technique according to randomization will be given after induction of general anesthesia Fentanyl boluses of 1 mcg/kg will be given in case of inadequate analgesia. Inadequate analgesia identified by 20% increase in the heart rate and/or systolic blood pressure from baseline measurement.

postoperative analgesia: regular paracetamol 1 g/6 hours (intravenously at first then orally once the oral feeding is resumed) and 75 mg diclofenac (intramuscularly at first then orally once the oral feeding is resumed).

If Numeric rating scale (NRS) is > 3 intravenous titration of 2 mg morphine is given slowly to be repeated after 30 minutes if pain persisted

ELIGIBILITY:
Inclusion Criteria:

* adult patients, undergoing open appendectomy.

Exclusion Criteria:

* American society of anesthesiologist-physical status >III,
* allergy to any of the study drugs,
* coagulopathy
* local infection,
* history of chronic pain or regular opioid use;
* inability to comprehend the Numeric Rating Scale (NRS),
* pregnant or lactating women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | from extubation until 24 hours postoperative
  mg

SECONDARY OUTCOMES:
numeric rating scale | AT 0.5, 2, 6, 12, and 24 hours postoperative.
  a scale of 0-10, where 0 means "no pain" and 10 means "worst imaginable pain"
quality of recovery | 24 hours after suregry
  assessed using Quality of recovery-15 (QOR-15); Consists of 15 items evaluating five dimensions of health: physical comfort, physical independence, psychological support, emotional state, and pain.
  Scoring Range: Each item is rated on an 11-point numerical scale (0 to 10). The total score ranges from 0 (extremely poor recovery) to 150 (excellent recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
data regarding this research will be available upon reasonable request from the PI